CLINICAL TRIAL: NCT02849418
Title: A Phase III Study to Evaluate the Efficacy and Safety of GSK1358820 (Botulinum Toxin Type A) in Patients With Urinary Incontinence Due to Neurogenic Detrusor Overactivity
Brief Title: Efficacy and Safety Study of GSK1358820 in Japanese Patients With Urinary Incontinence Due to Neurogenic Detrusor Overactivity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 204948
Record Dates: First submitted 2016-07-27; First posted 2016-07-29 (Estimated); Results first posted 2019-07-10 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Urinary Bladder, Overactive
Keywords: Botulinum toxin type A; Urinary Incontinence; Neurogenic Detrusor Overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK1358820 Injection 200 U (Experimental): Subjects will receive a single treatment with 200 U GSK1358820 injection (30 mL of study drug will be administered as 30 injections, each of 1.0 mL) in the detrusor of bladder, using cystoscopy and under local anesthesia. General anesthesia may be used excluding neuromuscular blocking agents. If the criteria for re-treatment between 12 to 36 weeks after first treatment are met, subjects will receive a second treatment with GSK1358820. Following this, subjects could receive another re-treatment up to 36 weeks after the first treatment, upon meeting the criteria, provided a minimum of 12 weeks elapse since previous treatment.
  Interventions: Drug: GSK1358820
- Placebo Injection (Placebo Comparator): Subjects will receive a single treatment with placebo (30 injections, each of 1 mL) in the detrusor of bladder, using cystoscopy and under local anesthesia. General anesthesia may be used excluding neuromuscular blocking agents. If the criteria for re-treatment between 12 to 36 weeks after first treatment are met, subjects will receive treatment with GSK1358820. Following this, subjects could receive another re-treatment up to 36 weeks after the first treatment, upon meeting the criteria, provided a minimum of 12 weeks elapse since previous treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK1358820 — GSK1358820 injection contains botulinum toxin type A (100 U), sodium chloride (0.9 milligrams [mg]), and human serum albumin (0.5 mg). The 30 mL of study drug will be administered as 30 injections each of 1.0 mL, evenly distributed at 30 sites in the detrusor muscle, spaced approximately 1 centimeter (cm) apart. The injection will be administered using cystoscopy and under local anesthesia. General anesthesia may be used excluding neuromuscular blocking agents.
  Arms: GSK1358820 Injection 200 U
Drug: Placebo — Placebo injection contains sodium chloride (0.9 milligrams [mg]); 30 mL of the injection will be injected at 30 sites in the detrusor muscle, spaced approximately 1 centimeter (cm) apart. The injection will be administered using cystoscopy and under local anesthesia. General anesthesia may be used excluding neuromuscular blocking agents
  Arms: Placebo Injection

SUMMARY:
This study will evaluate the efficacy and safety of GSK1358820 in Japanese patients with neurogenic detrusor overactivity (NDO) with urinary incontinence, whose symptoms have not been adequately managed with medications for urinary incontinence due to NDO.

This study consists of a screening phase up to 28 days followed by a double-blind Treatment phase 1 of 12 to 48 weeks wherein subjects will receive a single treatment of either GSK1358820 200 Units (U) injection or placebo injection. After the first treatment, subjects who meet the re-treatment criteria between 12 to 36 weeks can enter an open-label Treatment phase 2 to receive a second treatment with GSK1358820 200 U. Subjects will be permitted to receive re-treatment up to 2 times, and there should be a gap of minimum of 12 weeks since the previous treatment. The duration of overall treatment phases is 48 weeks. The total duration of participation for any subject will not exceed 52 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Aged >=20 years at the time of signing the informed consent
* Subject has urinary incontinence as a result of neurogenic detrusor overactivity for a period of at least 3 months prior to screening as a result of spinal cord injury or multiple sclerosis, determined by documented subject history. In addition:

  1. Spinal cord injury subjects must have a stable neurological injury level C5 or below occurring >=6 months prior to screening.
  2. Multiple sclerosis subjects must be clinically stable in the investigator's opinion, for >=3 months prior to screening and have an Expanded Disability Status Scale score <=6.5
* Subject has NDO for a period of at least 3 months prior to screening, determined by documented subject history. The presence of an involuntary detrusor contractions (IDC) must also be demonstrated during the urodynamic assessment during the screening period or Day 1 (prior to randomization).
* Subject has not been adequately managed with one or more medications (i.e., anticholinergics or beta-3 adrenergic receptor agonist) for treatment of urinary incontinence due to NDO . Not adequately managed is defined as:

An inadequate response after at least a 4-week period of medication(s) for urinary incontinence due to NDO on an optimized dose(s), i.e., subject is still incontinent despite medication(s) for urinary incontinence due to NDO, or Limiting side effects (i.e., condition that subject reduced dosage or discontinued the medication due to side effect) after at least a 2-week period of medication(s) for urinary incontinence due to NDO on an optimized dose(s)

* Subject has >=6 episodes of urinary incontinence, with no more than one urgency incontinence-free day in the 3-day subject bladder diary completed during the screening phase
* Subject currently uses or is willing to use clean intermittent catheterization (CIC) to empty the bladder (indwelling catheter is not permitted). Subjects currently on CIC should be willing to maintain a CIC schedule of at least 3 times per day throughout the study. Caregiver may perform CIC.
* Body weight >=40 kilogram (kg) at screening
* Males or females：

  1. Male subjects with female partners of child bearing potential must comply with the following contraception requirements from the time of first dose of study medication until the study exit:

     * Vasectomy with documentation of azoospermia.
     * Male condom plus partner use of one of following the contraceptive options:Intrauterine device or intrauterine system that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label; or oral contraceptive, either combined or progestogen alone These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception
  2. Female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine or serum human chorionic gonadotrophin [hCG] test), not lactating, and at least one of the following conditions applies:

     • Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation, Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, Hysterectomy, Documented Bilateral Oophorectomy.

     Postmenopausal defined as 12 months of spontaneous amenorrhea. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment.

     • Reproductive potential and agrees to follow one of the options listed below in the GlaxoSmithKline (GSK) Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from 30 days prior to the first dose of study medication and until the study exit. This list of highly effective methods (approved in Japan) is provided below, and it does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis: Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label; Oral Contraceptive, either combined or progestogen alone; Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

     These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Subject has given signed informed consent, including compliance with the requirements and restrictions listed in the consent form and in this protocol (e.g., complete bladder diaries and questionnaires, is able to collect volume voided per micturition measurements over a 24-hour period, and attend all study visits in the opinion of the investigator(or subinvestigator).

Exclusion Criteria:

* Subject has a history or evidence of any diseases, functional abnormalities or bladder surgery, other than NDO, that may have affected bladder function including but not limited to:

  1. Bladder stones (including bladder stone surgery) within 6 months prior to screening or confirmed occurrence of bladder stones at the screening phase
  2. Surgery (including minimally invasive surgery) within 1 year of screening for stress incontinence or pelvic organ prolapse
  3. Current use of an electrostimulation/neuromodulation device for treatment of urinary incontinence. Note: Use of any implantable device is prohibited within 4 weeks prior to initiation of Screening phase and throughout the study period. Use of any external device is discontinued at least 7 days prior to the start of the screening phase
  4. Current use of a baclofen pump
  5. History of interstitial cystitis, in the opinion of the investigator (or subinvestigator)
  6. Past or current evidence of hematuria due to urological/renal pathology or uninvestigated hematuria. Subjects with investigated hematuria may enter the study if urological/renal pathology has been ruled out to the satisfaction by the investigator (or subinvestigator)
  7. Past or current history of bladder cancer or other urothelial malignancy, positive result of urine cytology or uninvestigated suspicious urine cytology results at the Screening phase. Suspicious urine cytology abnormalities require that bladder cancer or other urothelial malignancy has been ruled out to the satisfaction of the investigator according to local site practice.
  8. An active genital infection, other than genital warts, either concurrently or within 4 weeks prior to Screening
  9. Male with previous or current diagnosis of prostate cancer or a prostate specific antigen (PSA) level of >10 nanogram (ng)/milliliter (mL) at Screening. Subjects with a PSA level of >= 4 ng/mL but <= 10 ng/mL must have prostate cancer ruled out to the satisfaction of the investigator (or subinvestigator) according to local site practice.
  10. Evidence of urethral and/or bladder outlet obstruction, in the opinion of the investigator (or subinvestigator)
* Subject has a serum creatinine level >2 times the upper limit of normal (ULN) at screening
* Alanine aminotransferase (ALT) > 2×ULN; and bilirubin > 1.5×ULN (isolated bilirubin >1.5×ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) at screening
* Subject has current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment). Notes:

  1. Stable chronic liver disease should generally be defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, oesophageal or gastric varices, or persistent jaundice, or cirrhosis
  2. Chronic stable hepatitis B and C (example, presence of hepatitis B surface antigen [HBsAg] or positive hepatitis C antibody [HCVAb] test result within 3 months prior to first dose of study treatment) are acceptable if subject otherwise meets entry criteria
* QTc >450 milliseconds (msec) or QTc >480 msec in subjects with Bundle Branch Block from the result of ECG at screening. Notes:

  1. The QTc is the QT interval corrected for heart rate according to Bazett's formula (QTcB), Fridericia's formula (QTcF), and/or another method, machine-read or manually over-read
  2. The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial
* Subject has hemophilia or other clotting factor deficiencies or disorders that cause bleeding diathesis
* Subject changes or initiates or discontinues anticholinergic, beta-3 adrenergic receptor agonist or any other medications or therapies to treat urinary incontinence due to NDO, within 6 days prior to the start of the screening phase
* Subject has been treated with any intravesical pharmacologic agent (e.g., capsaicin, resiniferatoxin) for urinary incontinence due to NDO within 12 months prior to initiation of Treatment phase 1 (Week 0)
* Subject has previous or current use of botulinum toxin therapy of any serotype for the treatment of any urological condition
* Subject has previous use within 12 weeks prior to initiation of Treatment phase 1 (Week 0) or current use of botulinum toxin therapy of any serotype for any non-urological condition or beauty care
* Subject has been immunized for botulinum toxin of any serotype
* Subject cannot withhold any antiplatelet or anticoagulant therapy or medications with anticoagulative effects for 3 days prior to initiation of Treatment phase 1 (Week 0). Some medications may need to be withheld for > 3 days, per clinical judgment of the investigator (or subinvestigator).
* Subject without a urinary tract infection (UTI) as determined from the urinalysis or urine culture and/or investigator opinion, has not initiated prophylactic antibiotic medication 1 to 3 days prior to the initiation of Treatment phase 1 (Week 0). Subject with a UTI as determined from the urinalysis or urine culture and/or investigator opinion, has not initiated antibiotic medication at least 5 days prior to the initiation of Treatment phase 1 (Week 0)
* Subject is symptomatic for UTI on day of treatment
* Subject has a history of sensitivity to any of the study medications, medications used in the study (including anesthesia), or their components or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* Subject has any medical condition that may put them at increased risk with exposure to GSK1358820 including diagnosed myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Females who are pregnant, nursing or planning a pregnancy during the study
* Subject has a post void residual urine volume above 200 mL for subjects who micturate or have a mixed catheterization/spontaneous micturition pattern. The post void residual measurement can be repeated once; the subject is to be excluded if the repeated measure is above 200 mL.
* Subject has a 24-hour total volume of urine voided >3000 mL of urine collected over 24 consecutive hours during the 3-day bladder diary collection period in the Screening phase
* Subject is currently participating in or has previously participated in another therapeutic study within 30 days prior to the start of the Screening phase
* Subject has any condition or situation which, in the investigator's (or sub-investigator's) opinion, puts the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (9):
- Japan (9):
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Yamanashi

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20849

REFERENCES:
- [Background] Honda M, Yokoyama O, Takahashi R, Matsuda T, Nakayama T, Mogi T. Botulinum toxin injections for Japanese patients with urinary incontinence caused by neurogenic detrusor overactivity: Clinical evaluation of onabotulinumtoxinA in a randomized, placebo-controlled, double-blind trial with an open-label extension. Int J Urol. 2021 Sep;28(9):906-912. doi: 10.1111/iju.14602. Epub 2021 Jun 1. PMID 34075630

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study evaluated the efficacy and safety of GSK1358820 (botulinum toxin type A) in participants with urinary incontinence due to neurogenic detrusor overactivity. This was a multicenter study conducted at 7 centers in Japan.
Pre-assignment Details: A total of 30 participants were screened of which 21 participants were randomized (11 participants in the GSK1358820 200 Unit [U] group and 10 participants in the placebo group).
Groups:
- Treatment Cycle 1: Placebo: Participants received a single (double-blind) treatment with Placebo (30 injections of 1.0 milliliter [mL] each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1).
- Treatment Cycle 1: GSK1358820 200U: Participants received a single (double-blind) dose of GSK1358820 200 U injections (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1).
- Treatment Cycle 2: Placebo / GSK1358820 200 U: Participants received a single (double-blind) treatment with Placebo (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received a single GSK1358820 200 U injection in the open-label Treatment Phase 2 (Treatment Cycle 2).
- Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U: Participants received a single (double-blind) dose of GSK1358820 (30 injections of 1.0 mL each) into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 200 U (open-label) in Treatment Phase 2 (Treatment Cycle 2).
- Treatment Cycle 3: Placebo / GSK1358820 200 U: Participants received a single (double-blind) treatment with Placebo (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants meeting the re-treatment criteria received a single GSK1358820 200 U injection in the open-label Treatment Phase 2 (Treatment Cycle 2) and further received re-treatment with GSK1358820 200 U in Treatment Phase 2 (Treatment Cycle 3).
- Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U: Participants received a single (double-blind) dose of GSK1358820 (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met re-treatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 200 U (open-label) in Treatment Phase 2 (Treatment Cycle 2) and further re-treatment with GSK1358820 200 U in Treatment Phase 2 (Treatment Cycle 3).
Period: Double-blinded (Up to 48 Weeks)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Started | 10 | 11 | 0 | 0 | 0 | 0
Completed | 10 | 11 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label(2nd Treatment-Week 12 to 48)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Started | 0 | 0 | 10 | 6 | 0 | 0
Completed | 0 | 0 | 10 | 6 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label(3rd Treatment-Week 12 to 48)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Started | 0 | 0 | 0 | 0 | 5 | 3
Completed | 0 | 0 | 0 | 0 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS1) Population comprised of all randomized participants who had at least 1 post-Baseline efficacy assessment.
Groups:
- Placebo: Participants received a single (double-blind) treatment with Placebo (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met retreatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 200 U (open-label) in Treatment Phase 2 until Week 36 after the first treatment and up to 2 times with an interval of at least 12 weeks between treatments.
- GSK1358820 200U: Participants received a single (double-blind) dose of GSK1358820 (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1). Participants who met retreatment criteria between 12 and 36 weeks after the first treatment received re-treatment with GSK1358820 200 U (open-label) in Treatment Phase 2 until Week 36 after the first treatment and up to 2 times with an interval of at least 12 weeks between treatments.
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK1358820 200U | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (18.29) | 50.9 (14.12) | 49.1 (15.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Japanese/East Asian (EA)/South EA Heritage | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes at Week 6
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Adjusted mean and standard error of adjusted mean has been reported.
Time Frame: Baseline (Pre-dose on Day 1) and Week 6 in Treatment Cycle 1
Population: FAS1 Population
Measure: Mean (Standard Error); unit: Episodes
Groups:
- Treatment Cycle 1: Placebo: Participants received a single (double-blind) treatment with Placebo (30 injections of 1.0 mL each) injected into the detrusor muscle of the bladder, using cystoscopy, and under local anesthesia in Treatment Phase 1 (Treatment Cycle 1).
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Episodes | -0.18 (0.957) | -3.20 (0.911)
Statistical Analysis 1: Comparison: Treatment Cycle 1: Placebo vs Treatment Cycle 1: GSK1358820 200U; Test type: Other; Mean Difference (Net) = -3.02, 95% CI 2-sided [-5.85 to -0.19] — The analysis method was mixed-model for repeated measures (MMRM) with treatment, visit, treatment-by-visit interaction, Baseline value, Baseline-by-visit interaction as fixed effects

2. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Maximum Cystometric Capacity (MCC) by Urodynamic Assessment at Week 6
Description: MCC was calculated by urodynamic assessment according to International Continence Society (ICS) standard guidelines. Baseline was the latest pre-dose assessment with a non-missing value. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1) and Week 6 in Treatment Cycle 1
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Milliliter | 62.05 (104.783) | 157.09 (161.159)

3. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Maximum Detrusor Pressure During the First Involuntary Detrusor Contraction (IDC) (PmaxIDC) by Urodynamic Assessment at Week 6
Description: PmaxIDC was calculated by urodynamic assessment according to ICS standard guidelines. Baseline was the latest pre-dose assessment with a non-missing value. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1) and Week 6 in Treatment Cycle 1
Population: FAS1 Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Centimeter of water (cmH2O)
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 8 | 6
Centimeter of water (cmH2O) | -0.005 (15.1414) | -21.000 (27.7705)

4. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Volume at First IDC (VPmaxIDC) by Urodynamic Assessment at Week 6
Description: VPmaxIDC was calculated by urodynamic assessment according to ICS standard guidelines. Baseline was the latest pre-dose assessment with a non-missing value. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1) and Week 6 in Treatment Cycle 1
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Milliliter | 67.7 (68.28) | 188.9 (157.43)

5. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Maximum Detrusor Pressure During the Storage Phase (PdetMax) by Urodynamic Assessment at Week 6
Description: PdetMax was calculated by urodynamic assessment according to ICS standard guidelines. Baseline was the latest pre-dose assessment with a non-missing value. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1) and Week 6 in Treatment Cycle 1
Population: FAS1 Population
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
cmH2O | -13.72 (29.141) | -31.18 (28.067)

6. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, Week 36, Week 42 and Week 48 in Treatment Cycle 1
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Episodes
  Week 2 | -0.90 (2.658) | -2.67 (2.530)
  Week 6 | -0.27 (3.321) | -3.12 (2.469)
  Week 12 | -0.40 (2.459) | -2.82 (2.518)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | -2.33 (0.943) | -3.46 (2.513)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | -2.50 (2.593) | -3.79 (2.295)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | -3.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -3.42 (2.195)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | -3.94 (2.832)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | -3.47 (2.181)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -3.80 (2.008)

7. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. FAS2 comprised all randomized participants who had at least 1 post-second treatment efficacy assessment after the second treatment.
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 18, Week 24, Week 30, and Week 36 in Treatment Cycle 2
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Episodes
  Week 0 | -0.33 (2.439) | -0.89 (1.026)
  Week 2 | -2.77 (2.735) | -1.06 (1.124)
  Week 6 | -3.17 (2.602) | -1.67 (0.919)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -2.56 (2.939) | -1.50 (0.983)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | -2.67 (2.041) | -1.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | -2.27 (3.157) | -1.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | -1.11 (3.657) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | 0.33 (4.243) |

8. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. FAS3 comprised all randomized participants who had at least 1 post-third treatment efficacy assessment after the third treatment.
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Episodes
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Episodes
  Week 0 | -1.47 (2.168) | -1.00 (0.577)
  Week 2 | -3.50 (1.732) | -1.44 (0.509)
  Week 6 | -3.87 (1.865) | -1.11 (0.839)
  Week 12 | -2.87 (2.219) | -1.56 (0.385)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -1.67 (0.943) | -1.50 (0.236)

9. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Percent Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data on the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Percent change
  Week 2 | -24.07 (38.593) | -59.07 (35.043)
  Week 6 | -10.58 (61.416) | -74.71 (36.316)
  Week 12 | -4.77 (60.523) | -67.64 (38.644)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | -42.31 (10.879) | -79.82 (24.361)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | -35.00 (21.213) | -91.07 (11.453)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | -38.46 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -79.99 (20.033)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | -78.83 (34.519)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | -78.70 (37.029)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -80.67 (26.390)

10. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Percent Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which has at least one valid diary day. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Percent change
  Week 0 | -2.77 (59.552) | -33.80 (37.522)
  Week 2 | -61.89 (45.317) | -46.30 (48.390)
  Week 6 | -67.47 (43.984) | -60.53 (32.686)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -43.22 (65.093) | -53.24 (36.701)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | -57.56 (36.509) | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | -33.05 (113.201) | -44.44 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | 1.28 (130.221) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | 52.56 (161.365) |

11. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Percent Change From Baseline in the Daily Average Number of Urinary Incontinence Episodes
Description: as for outcome 10
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Percent change
  Week 0 | -25.47 (47.584) | -28.70 (14.254)
  Week 2 | -73.55 (36.601) | -45.83 (18.162)
  Week 6 | -76.76 (33.447) | -43.29 (49.263)
  Week 12 | -51.18 (31.930) | -56.48 (38.922)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -21.29 (1.825) | -48.96 (25.043)

12. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in the Daily Average Number of Voids
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of void episodes. Data collected from a 24-hour period with less than 2 void episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which had at least one valid diary day assessment. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Voids
  Week 2 | -0.15 (1.253) | -0.79 (1.905)
  Week 6 | 0.10 (1.406) | -2.15 (3.354)
  Week 12 | 0.37 (1.869) | -2.24 (3.742)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | -0.83 (1.650) | -3.04 (3.827)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | -1.83 (0.707) | -2.88 (3.788)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | -3.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -2.54 (3.616)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | -2.83 (3.698)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | -2.20 (3.024)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -2.47 (3.548)

13. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in the Daily Average Number of Voids
Description: as for outcome 12
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Voids
  Week 0 | 0.10 (2.091) | -0.22 (1.601)
  Week 2 | -0.90 (1.343) | -0.72 (1.652)
  Week 6 | -1.33 (1.305) | -1.28 (1.819)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -0.96 (1.679) | 0.06 (1.902)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | 0.80 (0.869) | 2.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | 0.67 (1.247) | 0.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | 1.33 (2.000) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | 2.17 (1.650) |

14. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in the Daily Average Number of Voids
Description: as for outcome 12
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Voids
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Voids
  Week 0 | 0.27 (1.722) | 0.56 (1.018)
  Week 2 | -0.50 (1.908) | 0.22 (0.509)
  Week 6 | -0.47 (1.626) | 1.00 (1.155)
  Week 12 | -1.33 (2.789) | 0.11 (0.509)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -1.83 (3.064) | 0.17 (0.707)

15. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Percent Change From Baseline in the Daily Average Number of Voids
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of void episodes. Data collected from a 24-hour period with less than 2 void episodes (i.e., an invalid diary day) were set to missing. Baseline was defined as the latest pre-dose 3-day diary which had at least one valid diary day assessment. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Percent change
  Week 2 | -0.40 (14.219) | -5.62 (20.907)
  Week 6 | 1.10 (16.719) | -19.57 (26.762)
  Week 12 | 6.71 (20.180) | -19.59 (29.442)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | -7.01 (15.803) | -26.61 (27.085)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | -18.94 (3.214) | -24.02 (26.580)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | -27.27 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -19.61 (28.811)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | -20.61 (29.216)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | -14.15 (26.549)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -16.20 (27.755)

16. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Percent Change From Baseline in the Daily Average Number of Voids
Description: as for outcome 15
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Percent change
  Week 0 | 3.72 (22.732) | -1.67 (18.046)
  Week 2 | -8.40 (13.821) | -7.31 (18.173)
  Week 6 | -13.12 (11.015) | -16.44 (25.830)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -8.49 (16.813) | 1.97 (22.031)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | 10.33 (10.827) | 25.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | 8.18 (15.795) | 3.13 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | 17.53 (25.469) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | 28.33 (18.856) |

17. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Percent Change From Baseline in the Daily Average Number of Voids
Description: as for outcome 15
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Percent change
  Week 0 | 7.42 (15.640) | 8.79 (16.889)
  Week 2 | -0.38 (12.695) | 2.42 (6.042)
  Week 6 | -2.36 (16.615) | 12.95 (16.327)
  Week 12 | -7.14 (16.624) | 2.19 (8.054)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -6.82 (16.071) | 3.28 (11.071)

18. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Average Volume Voided Per Micturition
Description: The total volume voided was measured and recorded by participants over one 24-hour period during the 3-day bladder diary collection period. To perform this measurement, urine collection containers provided by the sponsor were used. The volume voided per void was determined by the sponsor from the total urine volume measured by the participants divided by the number of voids (excluding urinary incontinence episode). Baseline was defined as the latest pre-dose 3-day diary which had at least one valid diary day assessment. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Milliliter
  Week 2 | -3.68 (55.395) | 61.12 (50.470)
  Week 6 | 0.98 (86.368) | 107.53 (79.483)
  Week 12 | 6.85 (77.905) | 69.98 (64.010)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | 55.19 (44.989) | 84.11 (74.478)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | 53.65 (72.444) | 82.77 (61.992)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | 165.22 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 66.37 (48.478)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | 70.07 (26.988)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | 80.47 (42.477)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | 59.98 (6.616)

19. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 18
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Milliliter
  Week 0 | 7.83 (84.215) | 21.59 (38.130)
  Week 2 | 37.32 (78.467) | 76.01 (71.370)
  Week 6 | 54.67 (68.852) | 66.35 (76.721)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 51.28 (76.675) | 77.25 (68.182)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | -10.38 (60.659) | 60.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | 78.17 (96.434) | 57.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | 65.55 (196.119) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | -42.23 (114.691) |

20. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 18
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Milliliter
  Week 0 | -3.56 (78.698) | 68.62 (58.163)
  Week 2 | -17.78 (114.257) | 71.52 (51.555)
  Week 6 | -1.29 (116.143) | 59.27 (85.777)
  Week 12 | -0.96 (77.369) | 79.73 (26.835)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -0.72 (3.020) | 49.03 (21.572)

21. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Percent Change From Baseline in Average Volume Voided Per Micturition
Description: The total volume voided was measured and recorded by participants over one 24-hour period during the 3-day bladder diary collection period. To perform this measurement, urine collection containers provided by the sponsor were used. The volume voided per void was determined by the sponsor from the total urine volume measured by the participants divided by the number of voids (excluding urinary incontinence episode). Baseline was defined as the latest pre-dose 3-day diary which had at least one valid diary day assessment. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Percentage change from Baseline was calculated as post-dose visit value minus Baseline, divided by Baseline and multiplied by 100.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Percent change
  Week 2 | 4.14 (28.531) | 45.29 (38.910)
  Week 6 | 10.88 (53.306) | 76.99 (58.964)
  Week 12 | 12.56 (49.011) | 53.75 (53.789)
  Week 18: number analyzed (Participants) | 2 | 8
  Week 18 | 39.79 (36.933) | 71.03 (66.792)
  Week 24: number analyzed (Participants) | 2 | 8
  Week 24 | 40.43 (55.177) | 68.36 (54.836)
  Week 30: number analyzed (Participants) | 1 | 8
  Week 30 | 125.17 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 58.16 (51.203)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | 61.77 (46.781)
  Week 42: number analyzed (Participants) | 0 | 5
  Week 42 |  | 64.19 (34.387)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | 50.60 (24.805)

22. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Percent Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 21
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Percent change
  Week 0 | 13.72 (54.613) | 13.97 (26.244)
  Week 2 | 25.73 (51.374) | 48.31 (37.054)
  Week 6 | 37.32 (36.603) | 42.20 (50.162)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 30.25 (41.977) | 49.41 (50.110)
  Week 18: number analyzed (Participants) | 5 | 1
  Week 18 | -0.52 (25.276) | 42.19 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | 60.12 (78.234) | 39.86 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 30: number analyzed (Participants) | 3 | 0
  Week 30 | 68.58 (141.433) |
  Week 36: number analyzed (Participants) | 2 | 0
  Week 36 | -6.52 (52.333) |

23. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Percent Change From Baseline in Average Volume Voided Per Micturition
Description: as for outcome 21
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Percent change
  Week 0 | 1.72 (36.379) | 35.49 (21.018)
  Week 2 | -3.15 (50.796) | 43.15 (37.740)
  Week 6 | 3.41 (53.078) | 27.90 (39.969)
  Week 12 | 3.29 (33.790) | 46.12 (7.004)
  Week 18: number analyzed (Participants) | 2 | 2
  Week 18 | -0.27 (1.970) | 30.61 (23.706)

24. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Percentage of Participants Attaining 100 Percent (%), >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Percentage of participants attaining 100%, >=75% and >=50% reduction from Baseline in the daily average of urinary incontinence episodes in Treatment Cycle 1 have been presented.
Time Frame: as for outcome 6
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Percentage of participants
  Week 2, 100% | 0 | 18
  Week 2, >=75% | 0 | 36
  Week 2, >=50% | 40 | 73
  Week 6, 100% | 0 | 36
  Week 6, >=75% | 20 | 64
  Week 6, >=50% | 30 | 91
  Week 12, 100% | 0 | 27
  Week 12, >=75% | 0 | 64
  Week 12, >=50% | 20 | 73
  Week 18, 100%: number analyzed (Participants) | 2 | 8
  Week 18, 100% | 0 | 38
  Week 18, >=75%: number analyzed (Participants) | 2 | 8
  Week 18, >=75% | 0 | 63
  Week 18, >=50%: number analyzed (Participants) | 2 | 8
  Week 18, >=50% | 50 | 88
  Week 24, 100%: number analyzed (Participants) | 2 | 8
  Week 24, 100% | 0 | 38
  Week 24 >=75%: number analyzed (Participants) | 2 | 8
  Week 24 >=75% | 0 | 88
  Week 24 >=50%: number analyzed (Participants) | 2 | 8
  Week 24 >=50% | 50 | 100
  Week 30; 100%: number analyzed (Participants) | 1 | 8
  Week 30; 100% | 0 | 13
  Week 30; >=75%: number analyzed (Participants) | 1 | 8
  Week 30; >=75% | 0 | 75
  Week 30; >=50%: number analyzed (Participants) | 1 | 8
  Week 30; >=50% | 0 | 88
  Week 36; 100%: number analyzed (Participants) | 0 | 6
  Week 36; 100% |  | 50
  Week 36; >=75%: number analyzed (Participants) | 0 | 6
  Week 36; >=75% |  | 67
  Week 36; >=50%: number analyzed (Participants) | 0 | 6
  Week 36; >=50% |  | 83
  Week 42; 100%: number analyzed (Participants) | 0 | 5
  Week 42; 100% |  | 40
  Week 42; >=75%: number analyzed (Participants) | 0 | 5
  Week 42; >=75% |  | 80
  Week 42; >=50%: number analyzed (Participants) | 0 | 5
  Week 42; >=50% |  | 80
  Week 48; 100%: number analyzed (Participants) | 0 | 5
  Week 48; 100% |  | 20
  Week 48; >=75%: number analyzed (Participants) | 0 | 5
  Week 48; >=75% |  | 80
  Week 48; >=50%: number analyzed (Participants) | 0 | 5
  Week 48; >=50% |  | 80

25. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: Participants were instructed to enter data in the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Percentage of participants attaining 100%, >=75% and >=50% reduction from Baseline in the daily average of urinary incontinence episodes in Treatment Cycle 2 have been presented.
Time Frame: as for outcome 7
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Percentage of participants
  Week 0, 100% | 0 | 0
  Week 0, >=75% | 0 | 17
  Week 0, >=50% | 20 | 33
  Week 2, 100% | 20 | 33
  Week 2, >=75% | 60 | 33
  Week 2, >=50% | 80 | 50
  Week 6, 100% | 40 | 33
  Week 6, >=75% | 60 | 33
  Week 6, >=50% | 80 | 67
  Week 12, 100%: number analyzed (Participants) | 9 | 6
  Week 12, 100% | 33 | 17
  Week 12, >=75%: number analyzed (Participants) | 9 | 6
  Week 12, >=75% | 44 | 33
  Week 12, >=50%: number analyzed (Participants) | 9 | 6
  Week 12, >=50% | 67 | 50
  Week 18, 100%: number analyzed (Participants) | 5 | 1
  Week 18, 100% | 0 | 0
  Week 18, >=75%: number analyzed (Participants) | 5 | 1
  Week 18, >=75% | 40 | 0
  Week 18, >=50%: number analyzed (Participants) | 5 | 1
  Week 18, >=50% | 60 | 0
  Week 24, 100%: number analyzed (Participants) | 5 | 1
  Week 24, 100% | 40 | 0
  Week 24 >=75%: number analyzed (Participants) | 5 | 1
  Week 24 >=75% | 60 | 0
  Week 24 >=50%: number analyzed (Participants) | 5 | 1
  Week 24 >=50% | 80 | 0
  Week 30; 100%: number analyzed (Participants) | 3 | 0
  Week 30; 100% | 0 |
  Week 30; >=75%: number analyzed (Participants) | 3 | 0
  Week 30; >=75% | 33 |
  Week 30; >=50%: number analyzed (Participants) | 3 | 0
  Week 30; >=50% | 67 |
  Week 36; 100%: number analyzed (Participants) | 2 | 0
  Week 36; 100% | 0 |
  Week 36; >=75%: number analyzed (Participants) | 2 | 0
  Week 36; >=75% | 0 |
  Week 36; >=50%: number analyzed (Participants) | 2 | 0
  Week 36; >=50% | 50 |

26. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Percentage of Participants Attaining 100%, >=75% and >=50% Reduction From Baseline in the Daily Average of Urinary Incontinence Episodes
Description: Participants were instructed to enter data on the bladder diary over 3 consecutive days. For Baseline and post-treatment visits, analysis was based on the diary data collected during a 3-day interval for each visit. Each 3-day interval consisted of 3 consecutive 24-hour periods, with the first period starting from the time of the first urinary episode on the first of the 3 days. A valid diary day was defined as any of the three 24-hour periods with 2 or more any type of urinary incontinence episodes. Data collected from a 24-hour period with less than 2 urinary incontinence episodes (i.e., an invalid diary day) were set to missing. Percentage of participants attaining 100%, >=75% and >=50% reduction from Baseline in the daily average of urinary incontinence episodes in Treatment Cycle 3 have been presented.
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12 and Week 18 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Percentage of participants
  Week 0, 100% | 0 | 0
  Week 0, >=75% | 0 | 0
  Week 0, >=50% | 60 | 0
  Week 2, 100% | 20 | 0
  Week 2, >=75% | 80 | 0
  Week 2, >=50% | 80 | 33
  Week 6, 100% | 40 | 33
  Week 6, >=75% | 80 | 33
  Week 6, >=50% | 80 | 33
  Week 12, 100% | 20 | 33
  Week 12, >=75% | 20 | 33
  Week 12, >=50% | 40 | 33
  Week 18, 100%: number analyzed (Participants) | 2 | 2
  Week 18, 100% | 0 | 0
  Week 18, >=75%: number analyzed (Participants) | 2 | 2
  Week 18, >=75% | 0 | 0
  Week 18, >=50%: number analyzed (Participants) | 2 | 2
  Week 18, >=50% | 0 | 50

27. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Time to Qualification for Retreatment After First Treatment
Description: Participants can be considered for re-treatment beginning at the week 12 visit following the initial treatment or the week 12 visit following any re-treatment. Qualification criteria was; participants must have initiated request for re-treatment, participants experienced at least 4 episodes of urinary incontinence, with no more than one incontinence-free day, post-void residual (PVR) urine volume must have been <200 mL for participants who micturated or had a mixed catheterization / spontaneous micturition pattern, body weight >=40 kilogram; investigator deemed re-treatment appropriate. Time to the participant's first qualification for 2nd treatment from the day of 1st treatment was calculated as the earliest date when participants gave "Yes" response to the question of participants qualification for retreatment minus the day of first treatment plus 1.
Time Frame: Up to 36 Weeks in Treatment Cycle 1
Population: FAS1 Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Days | 85.0 [79.0 to 91.0] | 246.0 [84.0 to NA] — The data and very small number of participants did not allow calculation of the upper limit of 95% Confidence Interval.

28. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Time to Request for Retreatment After First Treatment
Description: The time taken by the participants to request re-treatment was reported. Time to the participant's first request for 2nd treatment from the day of 1st treatment was calculated as the earliest date when participants provided "Yes" response to the question of participants request for retreatment minus the day of first treatment plus 1.
Time Frame: Up to 36 Weeks in Treatment Cycle 1
Population: FAS1 Population
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Days | 84.5 [79.0 to 86.0] | 246.0 [84.0 to NA] — The data and very small number of participants did not allow calculation of the upper limit of 95% Confidence Interval.

29. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in King's Health Questionnaire (KHQ) Domain Score
Description: KHQ is a 21 item questionnaire, consisting of 9 domains:General health (GH) (1[Very good] to 5[Very poor]), Incontinence impact (Int Imp) (1[Not at all] to 4[A lot]), Role Limitations (RL) (1[Not at all] to 4[A lot]), Physical limitations (PL) (1[Not at all] to 4[A lot]), Social limitations (SL) (0[not applicable] to 4[A lot]), Personal relationships (PR) (0[Not applicable] to 4[A lot]), Emotions (1[Not at all] to 4[Very much]), Sleep or energy (S or E) (1[Never] to 4[All the time]) and Severity or Coping (S or C) (1[Never] to 4[All the time]). Domain score for GH was calculated as score of one item minus 1/4x100; Int Imp: score of one item minus 1/3x100; RL, PL, PR, S or E: summed scores of 2 items minus 2/6x100; SL, Emotions: summed scores of 3 items minus 3/9x100; S or C: summed scores of 5 items minus 5/15x100. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was any visit value minus Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 6, Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Scores on a scale
  General Health perception, Week 6 | 12.5 (13.18) | 6.8 (25.23)
  General Health Perception, Week 12 | 2.5 (18.45) | 9.1 (12.61)
  General Health Perception, Week 24: number analyzed (Participants) | 2 | 8
  General Health Perception, Week 24 | 12.5 (17.68) | 0.0 (13.36)
  General Health Perception, Week 36: number analyzed (Participants) | 1 | 6
  General Health Perception, Week 36 | 25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 16.7 (12.91)
  General Health Perception, Week 48: number analyzed (Participants) | 0 | 5
  General Health Perception, Week 48 |  | 15.0 (13.69)
  Incontinence impact, Week 6 | -6.67 (21.082) | -30.30 (43.345)
  Incontinence impact, Week 12 | -3.33 (33.148) | -30.30 (40.701)
  Incontinence impact, Week 24: number analyzed (Participants) | 2 | 8
  Incontinence impact, Week 24 | -16.67 (23.570) | -29.17 (33.034)
  Incontinence impact, Week 36: number analyzed (Participants) | 1 | 6
  Incontinence impact, Week 36 | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -38.89 (38.968)
  Incontinence impact, Week 48: number analyzed (Participants) | 0 | 5
  Incontinence impact, Week 48 |  | -26.67 (36.515)
  Role Limitations, Week 6 | -21.67 (20.861) | -12.12 (27.979)
  Role Limitations, Week 12 | -13.33 (29.187) | -12.12 (27.979)
  Role Limitations, Week 24: number analyzed (Participants) | 2 | 8
  Role Limitations, Week 24 | -16.67 (23.570) | -25.00 (30.861)
  Role Limitations, Week 36: number analyzed (Participants) | 1 | 6
  Role Limitations, Week 36 | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -27.78 (25.092)
  Role Limitations, Week 48: number analyzed (Participants) | 0 | 5
  Role Limitations, Week 48 |  | -10.00 (14.907)
  Physical Limitations, Week 6 | -20.00 (18.922) | -4.55 (44.778)
  Physical Limitations, Week 12 | -20.00 (24.595) | -15.15 (37.605)
  Physical Limitations, Week 24: number analyzed (Participants) | 2 | 8
  Physical Limitations, Week 24 | -25.00 (58.926) | -27.08 (34.431)
  Physical Limitations, Week 36: number analyzed (Participants) | 1 | 6
  Physical Limitations, Week 36 | -83.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -22.22 (32.773)
  Physical Limitations, Week 48: number analyzed (Participants) | 0 | 5
  Physical Limitations, Week 48 |  | -6.67 (9.129)
  Social Limitations, Week 6 | -16.67 (22.981) | -7.07 (47.212)
  Social Limitations, Week 12 | -24.44 (18.739) | -2.02 (41.520)
  Social Limitations, Week 24: number analyzed (Participants) | 2 | 8
  Social Limitations, Week 24 | -22.22 (15.713) | -25.00 (43.946)
  Social Limitations, Week 36: number analyzed (Participants) | 1 | 6
  Social Limitations, Week 36 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -11.11 (54.433)
  Social Limitations, Week 48: number analyzed (Participants) | 0 | 5
  Social Limitations, Week 48 |  | -0.00 (27.217)
  Personal Relationships, Week 6: number analyzed (Participants) | 8 | 8
  Personal Relationships, Week 6 | -10.42 (21.708) | 12.50 (38.576)
  Personal Relationships, Week 12: number analyzed (Participants) | 8 | 8
  Personal Relationships, Week 12 | 4.17 (45.207) | -4.17 (19.416)
  Personal Relationships, Week 24: number analyzed (Participants) | 1 | 7
  Personal Relationships, Week 24 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 2.38 (17.817)
  Personal Relationships, Week 36: number analyzed (Participants) | 1 | 5
  Personal Relationships, Week 36 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 6.67 (14.907)
  Personal Relationships, Week 48: number analyzed (Participants) | 0 | 4
  Personal Relationships, Week 48 |  | 8.33 (28.868)
  Emotions, Week 6 | 3.33 (27.242) | -9.09 (22.672)
  Emotions, Week 12 | -3.33 (24.595) | -8.08 (24.890)
  Emotions, Week 24: number analyzed (Participants) | 2 | 8
  Emotions, Week 24 | 0.00 (31.427) | -19.44 (23.570)
  Emotions, Week 36: number analyzed (Participants) | 1 | 6
  Emotions, Week 36 | 11.11 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -16.67 (29.606)
  Emotions, Week 48: number analyzed (Participants) | 0 | 5
  Emotions, Week 48 |  | -17.78 (18.592)
  Sleep/energy, Week 6 | -10.00 (23.831) | -7.58 (36.027)
  Sleep/energy, Week 12 | -11.67 (20.861) | -9.09 (35.248)
  Sleep/energy, Week 24: number analyzed (Participants) | 2 | 8
  Sleep/energy, Week 24 | 8.33 (11.785) | -18.75 (35.003)
  Sleep/energy, Week 36: number analyzed (Participants) | 1 | 6
  Sleep/energy, Week 36 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -16.67 (27.889)
  Sleep/energy, Week 48: number analyzed (Participants) | 0 | 5
  Sleep/energy, Week 48 |  | -0.00 (23.570)
  Severity/Coping measures, Week 6 | -9.33 (8.999) | -10.30 (20.519)
  Severity/Coping measures, Week 12 | -14.00 (15.854) | -14.55 (18.355)
  Severity/Coping measures, Week 24: number analyzed (Participants) | 2 | 8
  Severity/Coping measures, Week 24 | -6.67 (18.856) | -15.83 (23.077)
  Severity/Coping measures, Week 36: number analyzed (Participants) | 1 | 6
  Severity/Coping measures, Week 36 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -15.56 (17.213)
  Severity/Coping measures, Week 48: number analyzed (Participants) | 0 | 5
  Severity/Coping measures, Week 48 |  | -6.67 (13.333)

30. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in KHQ Domain Score
Description: KHQ is a 21 item questionnaire, consisting of 9 domains: GH (1[Very good] to 5[Very poor]), Int Imp (1[Not at all] to 4[A lot]), RL (1[Not at all] to 4[A lot]), PL (1[Not at all] to 4[A lot]), SL (0[not applicable] to 4[A lot]), PR (0[Not applicable] to 4[A lot]), Emotions (1[Not at all] to 4[Very much]), S or E (1[Never] to 4[All the time]) and S or C (1[Never] to 4[All the time]). Domain score for GH was calculated as score of one item minus 1/4x100; Int Imp: score of one item minus 1/3x100; RL, PL, PR, S or E: summed scores of 2 items minus 2/6x100; SL, Emotions: summed scores of 3 items minus 3/9x100; S or C: summed scores of 5 items minus 5/15x100. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was any visit value minus Baseline value.
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 6, Week 12, Week 24, and Week 36 in Treatment Cycle 2
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Scores on a scale
  General Health perception, Week 0 | 2.5 (18.45) | 12.5 (20.92)
  General Health perception, Week 6 | 5.0 (15.81) | 4.2 (18.82)
  General Health Perception, Week 12: number analyzed (Participants) | 9 | 6
  General Health Perception, Week 12 | 5.6 (20.83) | 12.5 (34.46)
  General Health Perception, Week 24: number analyzed (Participants) | 5 | 1
  General Health Perception, Week 24 | 10.0 (13.69) | -25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  General Health Perception, Week 36: number analyzed (Participants) | 3 | 0
  General Health Perception, Week 36 | 8.3 (14.43) |
  Incontinence Impact; Week 0 | -6.67 (34.427) | -16.67 (34.960)
  Incontinence Impact; Week 6 | -26.67 (40.976) | -33.33 (47.140)
  Incontinence Impact; Week 12: number analyzed (Participants) | 9 | 6
  Incontinence Impact; Week 12 | -25.93 (27.778) | -33.33 (47.140)
  Incontinence Impact; Week 24: number analyzed (Participants) | 5 | 1
  Incontinence Impact; Week 24 | -33.33 (40.825) | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Incontinence Impact; Week 36: number analyzed (Participants) | 3 | 0
  Incontinence Impact; Week 36 | -33.33 (33.333) |
  Role Limitations; Week 0 | -13.33 (29.187) | 2.78 (35.616)
  Role Limitations; Week 6 | -36.67 (36.683) | -5.56 (37.515)
  Role Limitations; Week 12: number analyzed (Participants) | 9 | 6
  Role Limitations; Week 12 | -37.04 (40.635) | 0.00 (38.006)
  Role Limitations; Week 24: number analyzed (Participants) | 5 | 1
  Role Limitations; Week 24 | -43.33 (34.561) | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Role Limitations; Week 36: number analyzed (Participants) | 3 | 0
  Role Limitations; Week 36 | -27.78 (25.459) |
  Physical Limitations; Week 0 | -21.67 (28.382) | 2.78 (41.388)
  Physical Limitations; Week 6 | -38.33 (29.450) | 0.00 (55.777)
  Physical Limitations; Week 12: number analyzed (Participants) | 9 | 6
  Physical Limitations; Week 12 | -40.74 (36.430) | -5.56 (51.280)
  Physical Limitations; Week 24: number analyzed (Participants) | 5 | 1
  Physical Limitations; Week 24 | -26.67 (30.277) | 16.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Physical Limitations; Week 36: number analyzed (Participants) | 3 | 0
  Physical Limitations; Week 36 | -38.89 (25.459) |
  Social Limitations; Week 0 | -21.11 (19.209) | 3.70 (58.654)
  Social Limitations; Week 6 | -35.56 (35.058) | -2.78 (57.922)
  Social Limitations; Week 12: number analyzed (Participants) | 9 | 6
  Social Limitations; Week 12 | -44.44 (24.845) | -8.33 (57.494)
  Social Limitations; Week 24: number analyzed (Participants) | 5 | 1
  Social Limitations; Week 24 | -44.44 (28.328) | 33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Social Limitations; Week 36: number analyzed (Participants) | 3 | 0
  Social Limitations; Week 36 | -37.04 (46.259) |
  Personal Relationships; Week 0: number analyzed (Participants) | 8 | 3
  Personal Relationships; Week 0 | 4.17 (45.207) | 5.56 (25.459)
  Personal Relationships; Week 6: number analyzed (Participants) | 8 | 3
  Personal Relationships; Week 6 | -20.83 (50.198) | 27.78 (63.099)
  Personal Relationships; Week 12: number analyzed (Participants) | 7 | 3
  Personal Relationships; Week 12 | -14.29 (45.571) | 22.22 (67.358)
  Personal Relationships; Week 24: number analyzed (Participants) | 4 | 1
  Personal Relationships; Week 24 | -16.67 (59.317) | 66.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Personal Relationships; Week 36: number analyzed (Participants) | 3 | 0
  Personal Relationships; Week 36 | -22.22 (38.490) |
  Emotions; Week 0 | -3.33 (22.253) | -3.70 (25.010)
  Emotions; Week 6 | -16.67 (35.234) | -5.56 (38.968)
  Emotions; Week 12: number analyzed (Participants) | 9 | 6
  Emotions; Week 12 | -9.88 (35.765) | -7.41 (38.915)
  Emotions; Week 24: number analyzed (Participants) | 5 | 1
  Emotions; Week 24 | -24.44 (39.597) | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Emotions; Week 36: number analyzed (Participants) | 3 | 0
  Emotions; Week 36 | -3.70 (39.021) |
  Sleep/Energy; Week 0 | -10.00 (21.082) | -0.00 (36.515)
  Sleep/Energy; Week 6 | -23.33 (21.082) | -5.56 (29.187)
  Sleep/Energy; Week 12: number analyzed (Participants) | 9 | 6
  Sleep/Energy; Week 12 | -16.67 (16.667) | -16.67 (34.960)
  Sleep/Energy; Week 24: number analyzed (Participants) | 5 | 1
  Sleep/Energy; Week 24 | -20.00 (27.386) | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Sleep/Energy; Week 36: number analyzed (Participants) | 3 | 0
  Sleep/Energy; Week 36 | 0.00 (16.667) |
  Severity/Coping Measures; Week 0 | -15.33 (13.717) | -12.22 (19.513)
  Severity/Coping Measures; Week 6 | -25.33 (23.476) | -11.11 (22.178)
  Severity/Coping Measures; Week 12: number analyzed (Participants) | 9 | 6
  Severity/Coping Measures; Week 12 | -25.93 (25.483) | -11.11 (22.965)
  Severity/Coping Measures; Week 24: number analyzed (Participants) | 5 | 1
  Severity/Coping Measures; Week 24 | -32.00 (21.807) | -33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Severity/Coping Measures; Week 36: number analyzed (Participants) | 3 | 0
  Severity/Coping Measures; Week 36 | -24.44 (20.367) |

31. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in KHQ Domain Score
Description: as for outcome 30
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 6, Week 12 and Week 24 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Scores on a scale
  General Health perception, Week 0 | 5.0 (20.92) | -16.7 (14.43)
  General Health perception, Week 6 | 5.0 (20.92) | -8.3 (14.43)
  General Health Perception, Week 12 | 10.0 (13.69) | -8.3 (14.43)
  General Health Perception, Week 24: number analyzed (Participants) | 1 | 0
  General Health Perception, Week 24 | 25.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Incontinence Impact; Week 0 | -20.00 (29.814) | -33.33 (0.000)
  Incontinence Impact; Week 6 | -40.00 (27.889) | -11.11 (38.490)
  Incontinence Impact; Week 12 | -20.00 (29.814) | -22.22 (19.245)
  Incontinence Impact; Week 24: number analyzed (Participants) | 1 | 0
  Incontinence Impact; Week 24 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Role Limitations; Week 0 | -30.00 (29.814) | 5.56 (9.623)
  Role Limitations; Week 6 | -50.00 (35.355) | -5.56 (25.459)
  Role Limitations; Week 12 | -33.33 (33.333) | 5.56 (41.944)
  Role Limitations; Week 24: number analyzed (Participants) | 1 | 0
  Role Limitations; Week 24 | 0.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Physical Limitations; Week 0 | -30.00 (21.731) | 16.67 (0.000)
  Physical Limitations; Week 6 | -43.33 (32.489) | 11.11 (9.623)
  Physical Limitations; Week 12 | -36.67 (27.386) | 16.67 (33.333)
  Physical Limitations; Week 24: number analyzed (Participants) | 1 | 0
  Physical Limitations; Week 24 | -16.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Social Limitations; Week 0 | -37.78 (23.040) | 9.26 (25.051)
  Social Limitations; Week 6 | -46.67 (24.088) | 7.41 (39.021)
  Social Limitations; Week 12 | -40.00 (21.660) | 18.52 (51.620)
  Social Limitations; Week 24: number analyzed (Participants) | 1 | 0
  Social Limitations; Week 24 | -11.11 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Personal Relationships; Week 0: number analyzed (Participants) | 4 | 1
  Personal Relationships; Week 0 | -12.50 (45.896) | 66.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Personal Relationships; Week 6: number analyzed (Participants) | 3 | 1
  Personal Relationships; Week 6 | -33.33 (66.667) | 66.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Personal Relationships; Week 12: number analyzed (Participants) | 4 | 1
  Personal Relationships; Week 12 | -16.67 (43.033) | 100.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Personal Relationships; Week 24: number analyzed (Participants) | 1 | 0
  Personal Relationships; Week 24 | 33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Emotions; Week 0 | -8.89 (30.832) | 7.41 (39.021)
  Emotions; Week 6 | -20.00 (30.832) | 7.41 (16.973)
  Emotions; Week 12 | -15.56 (26.759) | 7.41 (16.973)
  Emotions; Week 24: number analyzed (Participants) | 1 | 0
  Emotions; Week 24 | 22.22 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Sleep/Energy; Week 0 | -16.67 (16.667) | -5.56 (25.459)
  Sleep/Energy; Week 6 | -30.00 (13.944) | -5.56 (25.459)
  Sleep/Energy; Week 12 | -20.00 (13.944) | 0.00 (16.667)
  Sleep/Energy; Week 24: number analyzed (Participants) | 1 | 0
  Sleep/Energy; Week 24 | 33.33 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Severity/Coping Measures; Week 0 | -22.67 (12.111) | -4.44 (26.943)
  Severity/Coping Measures; Week 6 | -22.67 (13.824) | 4.44 (16.777)
  Severity/Coping Measures; Week 12 | -24.00 (12.996) | 0.00 (11.547)
  Severity/Coping Measures; Week 24: number analyzed (Participants) | 1 | 0
  Severity/Coping Measures; Week 24 | -26.67 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |

32. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Percentage of Participants With Positive Response on Treatment Benefit Scale (TBS)
Description: TBS consisted of 4 answers to 1 question, to which participants had to answer considering their current condition (urinary problems, urinary incontinence) compared to their condition before receiving any study treatment in the trial. Responses for questions were coded as 1 to 4 where 1 - Greatly improved, 2 - Improved, 3 - Not changed and 4 - Worsened. The answers of 1 - Greatly improved or 2 - Improved were regarded as positive response. Other answers including missing data were regarded as NO positive response.
Time Frame: Week 2, Week 6 , Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: FAS1 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Percentage of participants
  Week 2 | 10 | 55
  Week 6 | 20 | 91
  Week 12 | 30 | 73
  Week 24: number analyzed (Participants) | 1 | 8
  Week 24 | 0 | 100
  Week 36: number analyzed (Participants) | 1 | 6
  Week 36 | 0 | 100
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | 100

33. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Percentage of Participants With Positive Response on TBS
Description: as for outcome 32
Time Frame: Week 0, Week 2, Week 6, Week 12, Week 24, and Week 36 in Treatment Cycle 2
Population: FAS2 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Percentage of participants
  Week 0 | 30 | 33
  Week 2 | 70 | 67
  Week 6 | 80 | 83
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | 67 | 67
  Week 24: number analyzed (Participants) | 5 | 1
  Week 24 | 80 | 100
  Week 36: number analyzed (Participants) | 3 | 0
  Week 36 | 67 |

34. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Percentage of Participants With Positive Response on TBS
Description: as for outcome 32
Time Frame: Week 0, Week 2, Week 6, Week 12, and Week 24 in Treatment Cycle 3
Population: FAS3 Population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Percentage of participants
  Week 0 | 40 | 33
  Week 2 | 100 | 33
  Week 6 | 80 | 67
  Week 12 | 60 | 67
  Week 24: number analyzed (Participants) | 1 | 0
  Week 24 | 0 |

35. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Serious Adverse Events (SAEs) and Non-SAE
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety for double blind phase (SPDB) Population comprised of all participants who received at least one dose of study treatment.
Time Frame: Up to Week 48 in Treatment Cycle 1
Population: SPDB Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants
  SAEs | 1 | 1
  Non-SAEs | 5 | 8

36. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With SAEs and Non-SAEs: Placebo/GSK1358820 200 U
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety population 1 comprised of all participants who received at least one dose of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 10
Participants
  SAEs | 1
  Non-SAEs | 5

37. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With SAEs and Non-SAEs: GSK1358820 200 U / GSK1358820 200 U
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety Population 2 comprised of all participants who received at least two doses of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 6
Participants
  SAEs | 0
  Non-SAEs | 5

38. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With SAEs and Non-SAEs: Placebo / GSK1358820 200 U
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 5
Participants
  SAEs | 0
  Non-SAEs | 4

39. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With SAEs and Non-SAEs: GSK1358820 200 U / GSK1358820 200 U
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety Population 3 comprised of all participants who received three doses of GSK1358820.
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 3
Participants
  SAEs | 0
  Non-SAEs | 3

40. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Vital sign parameter SBP and DBP were measured in seated position after 5 minutes rest. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Millimeters of mercury
  SBP, Week 2 | 0.0 (16.31) | 7.3 (11.24)
  SBP, Week 6 | 1.9 (11.87) | 7.4 (14.60)
  SBP, Week 12 | 1.4 (13.94) | 6.2 (20.76)
  SBP, Week 24: number analyzed (Participants) | 1 | 8
  SBP, Week 24 | -15.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 11.6 (12.87)
  SBP, Week 36: number analyzed (Participants) | 0 | 6
  SBP, Week 36 |  | 2.7 (9.71)
  SBP, Week 48: number analyzed (Participants) | 0 | 5
  SBP, Week 48 |  | 7.4 (16.58)
  DBP, Week 2 | -1.8 (9.15) | 1.5 (9.77)
  DBP, Week 6 | 1.7 (8.78) | 4.6 (9.20)
  DBP, Week 12 | -0.4 (8.10) | 1.7 (12.45)
  DBP, Week 24: number analyzed (Participants) | 1 | 8
  DBP, Week 24 | -9.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 3.3 (8.80)
  DBP, Week 36: number analyzed (Participants) | 0 | 6
  DBP, Week 36 |  | 3.2 (5.15)
  DBP, Week 48: number analyzed (Participants) | 0 | 5
  DBP, Week 48 |  | 1.6 (6.91)

41. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in SBP and DBP
Description: as for outcome 40
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, Week 24 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Millimeters of mercury
  SBP, Week 0 | 3.3 (9.57) | 0.3 (8.19)
  SBP, Week 2 | -2.3 (16.64) | 8.2 (8.95)
  SBP, Week 6 | 2.6 (12.52) | 12.3 (8.09)
  SBP, Week 12: number analyzed (Participants) | 9 | 6
  SBP, Week 12 | -1.2 (12.71) | 6.0 (2.76)
  SBP, Week 24: number analyzed (Participants) | 4 | 1
  SBP, Week 24 | 3.5 (15.26) | -1.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  SBP, Week 48: number analyzed (Participants) | 5 | 3
  SBP, Week 48 | -0.2 (13.85) | 16.0 (12.17)
  DBP, Week 0 | -0.4 (10.70) | -1.3 (7.26)
  DBP, Week 2 | -3.5 (12.55) | 4.3 (10.61)
  DBP, Week 6 | 1.0 (8.25) | 4.2 (10.76)
  DBP, Week 12: number analyzed (Participants) | 9 | 6
  DBP, Week 12 | -4.6 (7.73) | 5.2 (7.44)
  DBP, Week 24: number analyzed (Participants) | 4 | 1
  DBP, Week 24 | 4.5 (9.95) | 6.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  DBP, Week 48: number analyzed (Participants) | 5 | 3
  DBP, Week 48 | 3.8 (10.38) | 11.3 (10.07)

42. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in SBP and DBP
Description: as for outcome 40
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 0, Week 2, Week 6, Week 12, and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Millimeters of mercury
  SBP, Week 0 | -5.0 (5.87) | 14.7 (8.50)
  SBP, Week 2 | 2.6 (13.22) | 8.3 (6.66)
  SBP, Week 6 | 1.8 (9.55) | 5.0 (6.08)
  SBP, Week 12: number analyzed (Participants) | 4 | 2
  SBP, Week 12 | 4.3 (11.98) | 2.5 (3.54)
  SBP, Week 48 | 6.0 (3.74) | 5.7 (15.50)
  DBP, Week 0 | -1.4 (4.22) | 1.3 (3.21)
  DBP, Week 2 | -1.0 (11.25) | 2.0 (12.49)
  DBP, Week 6 | -0.6 (8.32) | 6.3 (6.66)
  DBP, Week 12: number analyzed (Participants) | 4 | 2
  DBP, Week 12 | -4.5 (5.00) | 3.5 (0.71)
  DBP, Week 48 | -2.4 (5.86) | 4.0 (15.52)

43. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Heart Rate
Description: Vital sign parameter heart rate was measured in seated position after 5 minutes rest. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Beats per minute
  Week 2 | -1.3 (14.28) | -1.0 (10.80)
  Week 6 | 1.7 (12.64) | 4.5 (15.21)
  Week 12 | -1.4 (9.96) | 3.1 (6.01)
  Week 24: number analyzed (Participants) | 1 | 8
  Week 24 | -10.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -9.3 (9.79)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | 0.2 (12.86)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -13.0 (7.48)

44. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Heart Rate
Description: as for outcome 43
Time Frame: as for outcome 41
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Beats per minute
  Week 0 | 3.7 (12.57) | -3.5 (13.47)
  Week 2 | 0.1 (15.21) | 0.5 (13.87)
  Week 6 | 0.7 (16.75) | 2.2 (11.97)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -2.9 (16.59) | -1.8 (14.86)
  Week 24: number analyzed (Participants) | 4 | 1
  Week 24 | -5.3 (14.86) | 26.0 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 48: number analyzed (Participants) | 5 | 3
  Week 48 | -8.6 (7.83) | 1.3 (1.53)

45. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Heart Rate
Description: as for outcome 43
Time Frame: as for outcome 42
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Beats per minute
  Week 0 | 8.4 (12.90) | -5.0 (8.89)
  Week 2 | 5.4 (15.71) | -3.7 (23.71)
  Week 6 | 10.8 (19.07) | -7.0 (10.54)
  Week 12: number analyzed (Participants) | 4 | 2
  Week 12 | 8.5 (10.63) | -4.0 (8.49)
  Week 48 | 13.8 (12.62) | 2.7 (16.50)

46. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in Body Temperature
Description: Vital sign parameter temperature was measured in seated position after 5 minutes rest. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post-dose visit value from the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 24, Week 36 and Week 48 in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Degree Celsius
  Week 2 | 0.29 (0.438) | -0.06 (0.391)
  Week 6 | 0.05 (0.375) | -0.15 (0.401)
  Week 12 | 0.14 (0.460) | 0.03 (0.535)
  Week 24: number analyzed (Participants) | 1 | 8
  Week 24 | 0.30 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | -0.22 (0.471)
  Week 36: number analyzed (Participants) | 0 | 6
  Week 36 |  | -0.25 (0.550)
  Week 48: number analyzed (Participants) | 0 | 5
  Week 48 |  | -0.20 (0.400)

47. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in Body Temperature
Description: as for outcome 46
Time Frame: as for outcome 41
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Degree Celsius
  Week 0 | 0.16 (0.440) | -0.23 (0.186)
  Week 2 | 0.05 (0.536) | -0.07 (0.388)
  Week 6 | 0.15 (0.387) | 0.03 (0.344)
  Week 12: number analyzed (Participants) | 9 | 6
  Week 12 | -0.02 (0.315) | 0.02 (0.264)
  Week 24: number analyzed (Participants) | 4 | 1
  Week 24 | 0.53 (0.629) | 0.10 (NA) — Standard deviation could not be calculated as only one participant was analyzed.
  Week 48: number analyzed (Participants) | 5 | 3
  Week 48 | 0.26 (0.559) | -0.10 (0.173)

48. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in Body Temperature
Description: as for outcome 46
Time Frame: as for outcome 42
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Degree Celsius
  Week 0 | 0.06 (0.114) | -0.03 (0.153)
  Week 2 | 0.24 (0.270) | 0.23 (0.577)
  Week 6 | 0.20 (0.485) | 0.17 (0.351)
  Week 12: number analyzed (Participants) | 4 | 2
  Week 12 | 0.15 (0.370) | 0.10 (0.283)
  Week 48 | 0.08 (0.476) | 0.13 (0.666)

49. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Shift From Baseline in Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; Basophils, Eosinophils, Hemoglobin (Hb), Hematocrit (Hct), Lymphocytes (Lympho), Monocytes, Neutrophil bands (N bands), Total Neutrophils (T neutro), Platelet count (PC), Red Blood Cell (RBC) count, and White Blood Cell count (WBC). Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only categories with non-zero values have been presented.
Time Frame: Week 12, and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants
  Week 12: Basophils, Normal or no change | 10 | 11
  Week 48: Basophils, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48: Basophils, Normal or no change |  | 5
  Week 12: Eosinophils, Normal or no change | 9 | 11
  Week 12: Eosinophils, High | 1 | 0
  Week 48: Eosinophils, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48: Eosinophils, Normal or no change |  | 5
  Week12: Hb,Normal or no change | 10 | 11
  Week 48: Hb, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48: Hb, Normal or no change |  | 5
  Week 12:Hct, Normal or No change | 10 | 11
  Week 48: Hct, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48: Hct, Normal or no change |  | 5
  Week12:Lympho, Normal or no change | 10 | 10
  Week12:Lympho, High | 0 | 1
  Week48:Lympho, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48:Lympho, Normal or no change |  | 5
  Week 12:Monocytes, Normal or no change | 10 | 11
  Week48:Monocytes, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48:Monocytes, Normal or no change |  | 5
  Week 12:N bands, Normal or no change | 10 | 10
  Week 12:N bands, High | 0 | 1
  Week48: N bands, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48: N bands, Normal or no change |  | 5
  Week12:T neutro, Normal or no change | 10 | 11
  Week 48:T neutro, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:T neutro, Normal or no change |  | 5
  Week12:PC, Low | 0 | 1
  Week12:PC, Normal or no change | 9 | 10
  Week12:PC, High | 1 | 0
  Week48:PC, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48:PC, Normal or no change |  | 5
  Week12:RBC count, Normal or no change | 10 | 11
  Week48:RBC count, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48:RBC count, Normal or no change |  | 5
  Week12:WBC count, Low | 1 | 0
  Week12: WBC count, Normal to no change | 9 | 11
  Week48:WBC count, Normal or no change: number analyzed (Participants) | 0 | 5
  Week48:WBC count, Normal or no change |  | 5

50. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Shift From Baseline in Hematology Parameters
Description: Blood samples were collected from participants for analysis of following hematology parameters; Basophils, Eosinophils, Hb, Hct, Lympho, Monocytes, N bands, T neutro, PC, RBC count, and WBC. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, were recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only categories with non-zero values have been presented.
Time Frame: Week 12 and Week 48 (48 Weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 9 | 6
Participants
  Week 12: Basophils, Normal or no change | 9 | 6
  Week 48: Basophils, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48: Basophils, Normal or no change | 5 | 3
  Week 12: Eosinophils, Normal or no change | 9 | 6
  Week 48: Eosinophils, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48: Eosinophils, Normal or no change | 5 | 3
  Week 12: Hb,Low | 1 | 0
  Week12: Hb,Normal or no change | 8 | 6
  Week 48: Hb, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48: Hb, Normal or no change | 5 | 3
  Week 12:Hct, Normal or no change | 9 | 6
  Week 48: Hct, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48: Hct, Normal or no change | 5 | 3
  Week12:Lympho, Low | 1 | 0
  Week12:Lympho, Normal or no change | 8 | 6
  Week48:Lympho, Normal or No change: number analyzed (Participants) | 5 | 3
  Week48:Lympho, Normal or No change | 5 | 3
  Week 12:Monocytes, Normal or no change | 8 | 6
  Week 12:Monocytes, High | 1 | 0
  Week48:Monocytes, Normal or no change: number analyzed (Participants) | 5 | 3
  Week48:Monocytes, Normal or no change | 5 | 3
  Week 12:N bands, Normal or no change | 9 | 6
  Week48: N bands, Normal or no change: number analyzed (Participants) | 5 | 3
  Week48: N bands, Normal or no change | 5 | 3
  Week12:T neutro, Normal or no change | 7 | 6
  Week12:T neutro, High | 2 | 0
  Week 48:T neutro, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:T neutro, Normal or no change | 5 | 3
  Week12:PC, Normal or no change | 8 | 6
  Week12:PC, High | 1 | 0
  Week48:PC, Normal or No change: number analyzed (Participants) | 5 | 3
  Week48:PC, Normal or No change | 3 | 3
  Week48:PC, High: number analyzed (Participants) | 5 | 3
  Week48:PC, High | 2 | 0
  Week12:RBC count, Normal or no change | 9 | 6
  Week48:RBC count, Normal or No Change: number analyzed (Participants) | 5 | 3
  Week48:RBC count, Normal or No Change | 5 | 3
  Week12: WBC count, Low | 0 | 1
  Week12: WBC count, Normal to no change | 7 | 5
  Week12: WBC count, High | 2 | 0
  Week48:WBC count, Normal to no change: number analyzed (Participants) | 5 | 3
  Week48:WBC count, Normal to no change | 5 | 3

51. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Shift From Baseline in Hematology Parameters
Description: as for outcome 50
Time Frame: Week 12 and Week 48 (48 Weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Participants
  Week 12: Basophils, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12: Basophils, Normal or no change | 4 | 2
  Week 48: Basophils, Normal or no change | 5 | 3
  Week 12: Eosinophils, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12: Eosinophils, Normal or no change | 4 | 2
  Week 48: Eosinophils, Normal or no change | 5 | 3
  Week12: Hb,Normal or no change: number analyzed (Participants) | 4 | 2
  Week12: Hb,Normal or no change | 4 | 2
  Week48: Hb,Normal or no change | 4 | 3
  Week 48: Hb, High | 1 | 0
  Week 12:Hct, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Hct, Normal or no change | 4 | 2
  Week 48: Hct, Normal or no change | 5 | 3
  Week12:Lympho, Normal or no change: number analyzed (Participants) | 4 | 2
  Week12:Lympho, Normal or no change | 4 | 2
  Week48:Lympho, Normal or No change | 5 | 3
  Week 12:Monocytes, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Monocytes, Normal or no change | 4 | 2
  Week48:Monocytes, Normal or no change | 5 | 3
  Week 12:N bands, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:N bands, Normal or no change | 4 | 2
  Week48: N bands, Normal or no change | 5 | 3
  Week12:T neutro, Normal or no change: number analyzed (Participants) | 4 | 2
  Week12:T neutro, Normal or no change | 4 | 2
  Week 48:T neutro, Normal or no change | 5 | 3
  Week12:PC, Normal or no change: number analyzed (Participants) | 4 | 2
  Week12:PC, Normal or no change | 3 | 2
  Week12:PC, High: number analyzed (Participants) | 4 | 2
  Week12:PC, High | 1 | 0
  Week48:PC, Normal or No change | 4 | 3
  Week48:PC, High | 1 | 0
  Week12:RBC count, Normal or no change: number analyzed (Participants) | 4 | 2
  Week12:RBC count, Normal or no change | 4 | 2
  Week48:RBC count, Normal or No Change | 4 | 3
  Week48:RBC count, High | 1 | 0
  Week12: WBC count, Low: number analyzed (Participants) | 4 | 2
  Week12: WBC count, Low | 0 | 1
  Week12: WBC count, Normal to no change: number analyzed (Participants) | 4 | 2
  Week12: WBC count, Normal to no change | 4 | 1
  Week48: WBC count, Low | 0 | 1
  Week48: WBC count, Normal or no change | 4 | 2
  Week48:WBC count, High | 1 | 0

52. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Shift From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of following clinical chemistry parameters; Albumin, Alkaline Phosphatase (Alk Phosp), Alanine Amino Transferase (ALT), Aspartate Amino Transferase (AST), Direct Bilirubin (Bil), Total Bil, Calcium, Chloride, Creatinine, Glucose, Potassium, Sodium, Total Protein (T Protein), Urea/blood urea nitrogen (BUN) and Uric acid. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only categories with non-zero values have been presented.
Time Frame: Week 12 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants
  Week 12:Albumin, Low | 0 | 1
  Week 12:Albumin, Normal or no change | 10 | 10
  Week 48:Albumin, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Albumin, Normal or no change |  | 5
  Week 12:Alk phosp, Low | 0 | 1
  Week 12:Alk phosp, Normal or no change | 10 | 10
  Week 48:Alk phosp, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Alk phosp, Normal or no change |  | 5
  Week 12:ALT, Normal or no change | 10 | 11
  Week 48:ALT, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:ALT, Normal or no change |  | 5
  Week 12:AST, Normal or no change | 10 | 10
  Week 12:AST, High | 0 | 1
  Week 48:AST, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:AST, Normal or no change |  | 5
  Week 12:Direct Bil, Normal or no change | 10 | 10
  Week 12:Direct Bil, High | 0 | 1
  Week 48:Direct Bil, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Direct Bil, Normal or no change |  | 5
  Week 12:Total Bil, Normal or no change | 10 | 10
  Week 12:Total Bil, High | 0 | 1
  Week 48:Total Bil, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Total Bil, Normal or no change |  | 5
  Week 12:Calcium, Low | 0 | 1
  Week 12:Calcium, Normal or no change | 10 | 10
  Week 48:Calcium, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Calcium, Normal or no change |  | 5
  Week 12:Chloride, Normal or no change | 10 | 11
  Week 48:Chloride, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Chloride, Normal or no change |  | 5
  Week 12:Creatinine, Low | 1 | 0
  Week 12:Creatinine, Normal or no change | 9 | 10
  Week 12:Creatinine, High | 0 | 1
  Week 48:Creatinine, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Creatinine, Normal or no change |  | 5
  Week 12:Glucose, Normal or no change | 8 | 7
  Week 12:Glucose, High | 2 | 4
  Week 48:Glucose, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Glucose, Normal or no change |  | 5
  Week 12:Potassium, Normal or no change | 10 | 11
  Week 48:Potassium, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Potassium, Normal or no change |  | 5
  Week 12:Sodium, Normal or no change | 10 | 11
  Week 48:Sodium, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Sodium, Normal or no change |  | 5
  Week 12:T protein, Low | 0 | 1
  Week 12:T protein, Normal or no change | 10 | 10
  Week 48:T protein, Low: number analyzed (Participants) | 0 | 5
  Week 48:T protein, Low |  | 1
  Week 48:T protein, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:T protein, Normal or no change |  | 4
  Week 12:Urea/BUN, Normal or no change | 9 | 11
  Week 12:Urea/BUN, High | 1 | 0
  Week 48:Urea/BUN, Low: number analyzed (Participants) | 0 | 5
  Week 48:Urea/BUN, Low |  | 1
  Week 48:Urea/BUN, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Urea/BUN, Normal or no change |  | 4
  Week 12:Uric acid, Normal or no change | 9 | 11
  Week 12:Uric acid, High | 1 | 0
  Week 48:Uric acid, Normal or no change: number analyzed (Participants) | 0 | 5
  Week 48:Uric acid, Normal or no change |  | 5

53. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Shift From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for analysis of following clinical chemistry parameters; Albumin, Alk Phosp, ALT, AST, Direct Bil, Total Bil, Calcium, Chloride, Creatinine, Glucose, Potassium, Sodium, T Protein, Urea/BUN and Uric acid. Participants were counted in the worst case category that their value changes to (Low, Normal or High), unless there is no change in their category. Participants whose value category was unchanged (e.g. High to High) or whose value became normal, are recorded in the 'To Normal or No Change' category. Participants were counted twice if the participant had values that changed 'To Low' and 'To High', so the percentages may not add to 100 percent. Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Only categories with non-zero values have been presented.
Time Frame: Week 12 and Week 48 (48 Weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 9 | 6
Participants
  Week 12: Albumin, Normal or no change | 9 | 6
  Week 48:Albumin, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Albumin, Normal or no change | 5 | 3
  Week 12:Alk phosp, Normal or no change | 9 | 6
  Week 48:Alk phosp, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Alk phosp, Normal or no change | 4 | 3
  Week 48:Alk phosp, High: number analyzed (Participants) | 5 | 3
  Week 48:Alk phosp, High | 1 | 0
  Week 12:ALT, Normal or no change | 9 | 5
  Week 12:ALT, High | 0 | 1
  Week 48:ALT, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:ALT, Normal or no change | 5 | 3
  Week 12:AST, Normal or no change | 9 | 5
  Week 12:AST, High | 0 | 1
  Week 48:AST, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:AST, Normal or no change | 5 | 2
  Week 48:AST, High: number analyzed (Participants) | 5 | 3
  Week 48:AST, High | 0 | 1
  Week 12:Direct Bil, Normal or no change | 9 | 6
  Week 48:Direct Bil, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Direct Bil, Normal or no change | 5 | 3
  Week 12:Total Bil, Normal or no change | 9 | 6
  Week 48:Total Bil, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Total Bil, Normal or no change | 5 | 3
  Week 12:Calcium, Low | 0 | 1
  Week 12:Calcium, Normal or no change | 9 | 5
  Week 48:Calcium, Low: number analyzed (Participants) | 5 | 3
  Week 48:Calcium, Low | 0 | 1
  Week 48:Calcium, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Calcium, Normal or no change | 5 | 2
  Week 12:Chloride, Normal or no change | 9 | 6
  Week 48:Chloride, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Chloride, Normal or no change | 5 | 3
  Week 12:Creatinine, Low | 1 | 0
  Week 12:Creatinine, Normal or no change | 8 | 6
  Week 48:Creatinine, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Creatinine, Normal or no change | 5 | 3
  Week 12:Glucose, Normal or no change | 8 | 4
  Week 12:Glucose, High | 1 | 2
  Week 48:Glucose, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Glucose, Normal or no change | 4 | 2
  Week 48:Glucose, High: number analyzed (Participants) | 5 | 3
  Week 48:Glucose, High | 1 | 1
  Week 12:Potassium, Normal or no change | 9 | 6
  Week 48:Potassium, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Potassium, Normal or no change | 5 | 3
  Week 12:Sodium, Normal or no change | 9 | 6
  Week 48:Sodium, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Sodium, Normal or no change | 5 | 3
  Week 12:T protein, Normal or no change | 9 | 6
  Week 48:T protein, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:T protein, Normal or no change | 5 | 3
  Week 12:Urea/BUN, Normal or no change | 9 | 6
  Week 48:Urea/BUN, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Urea/BUN, Normal or no change | 5 | 3
  Week 12:Uric acid, Normal or no change | 7 | 6
  Week 12:Uric acid, High | 2 | 0
  Week 48:Uric acid, Normal or no change: number analyzed (Participants) | 5 | 3
  Week 48:Uric acid, Normal or no change | 4 | 3
  Week 48:Uric acid, High: number analyzed (Participants) | 5 | 3
  Week 48:Uric acid, High | 1 | 0

54. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Shift From Baseline in Clinical Chemistry Parameters
Description: as for outcome 53
Time Frame: Week 12 and Week 48 (48 Weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Participants
  Week 12:Albumin, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Albumin, Normal or no change | 4 | 2
  Week 48:Albumin, Normal or no change | 5 | 3
  Week 12:Alk phosp, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Alk phosp, Normal or no change | 4 | 2
  Week 48:Alk phosp, Normal or no change | 5 | 3
  Week 12:ALT, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:ALT, Normal or no change | 3 | 2
  Week 12:ALT, High: number analyzed (Participants) | 4 | 2
  Week 12:ALT, High | 1 | 0
  Week 48:ALT, Normal or no change | 4 | 3
  Week 48:ALT, High | 1 | 0
  Week 12:AST, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:AST, Normal or no change | 3 | 2
  Week 12:AST, High: number analyzed (Participants) | 4 | 2
  Week 12:AST, High | 1 | 0
  Week 48:AST, Normal or no change | 4 | 3
  Week 48:AST, High | 1 | 0
  Week 12:Direct Bil, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Direct Bil, Normal or no change | 4 | 2
  Week 48:Direct Bil, Normal or no change | 5 | 3
  Week 12:Total Bil, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Total Bil, Normal or no change | 4 | 2
  Week 48:Total Bil, Normal or no change | 5 | 3
  Week 12:Calcium, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Calcium, Normal or no change | 4 | 2
  Week 48:Calcium, Normal or no change | 5 | 3
  Week 12:Chloride, Low: number analyzed (Participants) | 4 | 2
  Week 12:Chloride, Low | 1 | 0
  Week 12:Chloride, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Chloride, Normal or no change | 3 | 2
  Week 48:Chloride, Low | 1 | 0
  Week 48:Chloride, Normal or no change | 4 | 3
  Week 12:Creatinine, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Creatinine, Normal or no change | 4 | 2
  Week 48:Creatinine, Low | 1 | 0
  Week 48:Creatinine, Normal or no change | 4 | 3
  Week 12:Glucose, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Glucose, Normal or no change | 3 | 2
  Week 12:Glucose, High: number analyzed (Participants) | 4 | 2
  Week 12:Glucose, High | 1 | 0
  Week 48:Glucose, Normal or no change | 4 | 3
  Week 48:Glucose, High | 1 | 0
  Week 12:Potassium, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Potassium, Normal or no change | 4 | 2
  Week 48:Potassium, Normal or no change | 5 | 3
  Week 12:Sodium, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Sodium, Normal or no change | 4 | 2
  Week 48:Sodium, Normal or no change | 5 | 3
  Week 12:T protein, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:T protein, Normal or no change | 3 | 2
  Week 12:T protein, High: number analyzed (Participants) | 4 | 2
  Week 12:T protein, High | 1 | 0
  Week 48:T protein, Normal or no change | 4 | 3
  Week 48:T protein | 1 | 0
  Week 12:Urea/BUN, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Urea/BUN, Normal or no change | 4 | 2
  Week 48:Urea/BUN, Low | 0 | 1
  Week 48:Urea/BUN, Normal or no change | 5 | 2
  Week 12:Uric acid, Low: number analyzed (Participants) | 4 | 2
  Week 12:Uric acid, Low | 1 | 0
  Week 12:Uric acid, Normal or no change: number analyzed (Participants) | 4 | 2
  Week 12:Uric acid, Normal or no change | 3 | 2
  Week 48:Uric acid, Normal or no change | 5 | 3

55. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Analysis
Description: Urinalysis parameters assessed were urine occult blood, urine protein. In this dipstick test, the level of occult blood and protein in urine samples was recorded as negative, trace, 1+, 2+, 3+ and 4+ (the plus sign increases with a higher level of occult blood or proteins in the urine: 1+=slightly positive, 2+=positive, 3+=high positive etc). Baseline is the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Number of participants with worst-case urinalysis results post-Baseline relative to Baseline by dipstick analysis have been presented.
Time Frame: Baseline (Pre-dose on Day 1) and up to Week 48 in Treatment Cycle 1
Population: SPDB Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants
  Occult blood, Any Increase | 3 | 6
  Occult blood, Increase to Trace | 2 | 1
  Occult blood, Increase to 1+ | 0 | 4
  Increase to 2+ | 0 | 0
  Increase to 3+ | 1 | 1
  Increase to 4+ | 0 | 0
  Protein, Any Increase | 2 | 2
  Protein, Increase to Trace | 1 | 1
  Protein, Increase to 1+ | 1 | 1
  Protein, Increase to 2+ | 0 | 0
  Protein, Increase to 3+ | 0 | 0
  Protein, Increase to 4+ | 0 | 0

56. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Analysis
Description: as for outcome 55
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1) and up to 48 weeks after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 10 | 6
Participants
  Occult blood, Any Increase | 2 | 2
  Occult blood, Increase to Trace | 0 | 1
  Occult blood, Increase to 1+ | 1 | 1
  Increase to 2+ | 1 | 0
  Increase to 3+ | 0 | 0
  Increase to 4+ | 0 | 0
  Protein, Any Increase | 1 | 0
  Protein, Increase to Trace | 0 | 0
  Protein, Increase to 1+ | 1 | 0
  Protein, Increase to 2+ | 0 | 0
  Protein, Increase to 3+ | 0 | 0
  Protein, Increase to 4+ | 0 | 0

57. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Worst-case Urinalysis Results Post-Baseline Relative to Baseline by Dipstick Analysis
Description: as for outcome 55
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1) and up to 48 weeks after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Participants
  Occult blood, Any Increase | 2 | 1
  Occult blood, Increase to Trace | 1 | 0
  Occult blood, Increase to 1+ | 0 | 0
  Increase to 2+ | 0 | 0
  Increase to 3+ | 1 | 1
  Increase to 4+ | 0 | 0
  Protein, Any Increase | 2 | 1
  Protein, Increase to Trace | 2 | 1
  Protein, Increase to 1+ | 0 | 0
  Protein, Increase to 2+ | 0 | 0
  Protein, Increase to 3+ | 0 | 0
  Protein, Increase to 4+ | 0 | 0

58. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Urinary Tract Infection (UTI)
Description: A urine culture and sensitivity test were performed when urinalysis results with a urine reagent strip are suggestive of a UTI (positive nitrites or leukocyte esterase). UTI was recorded as an AE, irrespective of symptoms when the result of urine culture was positive (with the presence of bacteriuria with >=10^5 Colony Forming Unit per milliliter (CFU/mL) and leukocyturia with >5 per high power field was noted. Number of participants with UTI undergoing urine culture and sensitivity analysis have been presented.
Time Frame: Up to Week 48 in Treatment Cycle 1
Population: SPDB Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants | 0 | 2

59. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With UTI: Placebo/GSK1358820 200 U
Description: A urine culture and sensitivity test were performed when urinalysis results with a urine reagent strip are suggestive of a UTI (positive nitrites or leukocyte esterase). UTI was recorded as an AE, irrespective of symptoms when the result of urine culture was positive (with the presence of bacteriuria with >=10^5 CFU/mL and leukocyturia with >5 per high power field was noted. Number of participants with UTI undergoing urine culture and sensitivity analysis have been presented.
Time Frame: Up to Week 48 after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 10
Participants | 3

60. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With UTI: GSK1358820 200 U/GSK1358820 200 U
Description: as for outcome 59
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 6
Participants | 1

61. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With UTI: Placebo/GSK1358820 200 U
Description: as for outcome 59
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 5
Participants | 2

62. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With UTI: GSK1358820 200 U/GSK1358820 200 U
Description: as for outcome 59
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 3
Participants | 2

63. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Change From Baseline in PVR Urine Volume
Description: PVR was measured in non-catheterizing participants, or those with mixed patterns (ie, they do both clean intermittent catheterization [CIC] and spontaneous voiding). PVR urine volume was assessed by ultrasound, bladder scan or catheterization after participants performed a voluntary void according to the study schedule. PVR urine volume could be assessed at any other time depending on clinical need. In case PVR urine volume indicated a clinically meaningful elevation, participants were asked to void once again (allowing the participants sufficient time to void) and the PVR urine volume was then reassessed. For participants who had a PVR urine volume measurement repeated, only the repeat value was recorded. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Pre-dose on Day 1), Week 2, Week 6, Week 12, Week 24, Week 36 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 3 | 3
Milliliter
  Week 2: number analyzed (Participants) | 2 | 3
  Week 2 | 6.25 (8.839) | 166.50 (244.340)
  Week 6 | 25.33 (22.143) | 87.00 (175.997)
  Week 12 | -30.73 (47.963) | 177.03 (245.670)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 24.00 (NA) — Standard deviation could not be calculated as only one participant was analyzed. | 208.85 (45.891)
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 206.65 (196.081)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 207.10 (231.648)

64. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in PVR Urine Volume: Placebo / GSK1358820 200 U
Description: PVR was measured in non-catheterizing participants, or those with mixed patterns (ie, they do both CIC and spontaneous voiding). PVR urine volume was assessed by ultrasound, bladder scan or catheterization after participants performed a voluntary void according to the study schedule. PVR urine volume could be assessed at any other time depending on clinical need. In case PVR urine volume indicated a clinically meaningful elevation, participants were asked to void once again (allowing the participants sufficient time to void) and the PVR urine volume was then reassessed. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 2, Week 6 and Week 12 (Study exit, Week 48 of Treatment Cycle 1) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Milliliter
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 2
Milliliter
  Week 2 | 46.5 [0 to 93]
  Week 6 | 42 [0 to 84]
  Week 12 | 1 [0 to 2]

65. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Change From Baseline in PVR Urine Volume: GSK1358820 200 U / GSK1358820 200 U
Description: PVR was measured in non-catheterizing participants, or those with mixed patterns (ie, they do both CIC and spontaneous voiding). PVR urine volume was assessed by ultrasound, bladder scan or catheterization after participants performed a voluntary void according to the study schedule. PVR urine volume could be assessed at any other time depending on clinical need. In case PVR urine volume indicated a clinically meaningful elevation, participants were asked to void once again (allowing the participants sufficient time to void) and the PVR urine volume was then reassessed. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. Individual participant data has been presented.
Time Frame: as for outcome 64
Population: Safety Population 2. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Milliliter
Arm/Group | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 1
Milliliter
  Participant 1: Week 2 | -129.8
  Participant 1: Week 6 | -129.8
  Participant 1: Week 12 | -144.8

66. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in PVR Urine Volume: Placebo / GSK1358820 200 U
Description: as for outcome 65
Time Frame: Baseline (Day 1, pre-dose of Treatment Cycle 1), Week 2, Week 6, Week 12 and Week 48 (study exit or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 2. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Milliliter
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 1
Milliliter
  Participant 1: Week 2 | 47
  Participant 1: Week 6 | 84
  Participant 1: Week 12 | 0
  Participant 1: Week 48 | 0

67. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Change From Baseline in PVR Urine Volume: GSK1358820 200 U / GSK1358820 200 U
Description: as for outcome 65
Time Frame: as for outcome 66
Population: Safety Population 3. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Milliliter
Arm/Group | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 1
Milliliter
  Participant 1: Week 2 | -129.8
  Participant 1: Week 6 | -134.8
  Participant 1: Week 12 | -12.5
  Participant 1: Week 48 | -90.8

68. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants Using CIC for Urinary Retention or Elevated PVR
Description: CIC was used to drain the bladder and manage urinary incontinence in participants who were not able to spontaneously void. Participants who had used CIC at least once after the first treatment with the reason for urinary retention or elevated PVR have been presented.
Time Frame: Up to Week 48 in Treatment Cycle 1
Population: SPDB Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants | 0 | 1

69. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: Placebo / GSK1358820 200 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 10
Participants | 0

70. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: GSK1358820 200 U / GSK1358820 200 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 6
Participants | 0

71. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: Placebo / GSK1358820 200 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 5
Participants | 0

72. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants Using CIC for Urinary Retention or Elevated PVR: GSK1358820 200 U / GSK1358820 200 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 3
Participants | 0

73. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Abnormal Findings in Kidney and Bladder Ultrasound Examination
Description: The kidney and bladder ultrasound study was performed according to the study schedule. In order to assess the presence of stones in the kidneys and bladder, an ultrasound of these structures (with the bladder at least half full) was performed. Participants were excluded from this study if the screening ultrasound demonstrated the presence of bladder stones. In the case of unclear findings in an ultrasound study, other diagnostic measures (e.g., x-ray) was required in order to confirm the presence of bladder stones. If a stone was detected in participants after the injection of the investigational product, the event was recorded as an adverse event.
Time Frame: Up to Week 48 in Treatment Cycle 1
Population: SPDB Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

74. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Abnormal Findings in Kidney and Bladder Ultrasound Examination: Placebo / GSK1358820 200 U
Description: as for outcome 73
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 10
Participants | 0

75. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With Abnormal Findings in Kidney and Bladder Ultrasound Examination: GSK1358820 200 U / GSK1358820 200 U
Description: as for outcome 73
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 6
Participants | 0

76. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Abnormal Findings in Kidney and Bladder Ultrasound Examination: Placebo / GSK1358820 200 U
Description: as for outcome 73
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U
Number analyzed (Participants) | 5
Participants | 0

77. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With Abnormal Findings in Kidney and Bladder Ultrasound Examination: GSK1358820 200 U / GSK1358820 200 U
Description: as for outcome 68
Time Frame: Up to 48 weeks after 1st treatment
Population: Safety Population 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 3
Participants | 0

78. Secondary Outcome: Treatment Phase 1 (Treatment Cycle 1)- Number of Participants With Abnormal Not Clinically Significant (A-NCS) and Abnormal Clinically Significant (A-CS) Electrocardiogram (ECG) Findings
Description: Single 12-lead ECGs were obtained at each timepoint during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT intervals. The findings from ECG were classified as A-NCS and A-CS. Number of participants with A-NCS and A-CS findings have been reported.
Time Frame: Baseline (Pre-dose on Day 1), Week 12 and Week 48 in Treatment Cycle 1
Population: SPDB Population. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U
Number analyzed (Participants) | 10 | 11
Participants
  Baseline: A-NCS | 1 | 0
  Baseline: A-CS | 0 | 0
  Week 12: A-NCS | 1 | 1
  Week 12: ACS | 0 | 0
  Week 48: A-NCS: number analyzed (Participants) | 0 | 5
  Week 48: A-NCS |  | 1
  Week 48: A-CS: number analyzed (Participants) | 0 | 5
  Week 48: A-CS |  | 0

79. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 2)- Number of Participants With A-NCS and A-CS ECG Findings
Description: Single 12-lead ECGs were obtained at each timepoint during the study using an ECG machine that automatically calculated the heart rate and measured PR, QRS, and QT. The findings from ECG were classified as A-NCS and A-CS. Number of participants with A-NCS and A-CS findings have been reported.
Time Frame: Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 2
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 9 | 6
Participants
  Week 12: A-NCS | 1 | 0
  Week 12: A-CS | 0 | 0
  Week 48: A-NCS: number analyzed (Participants) | 5 | 3
  Week 48: A-NCS | 0 | 0
  Week 48: A-CS: number analyzed (Participants) | 5 | 3
  Week 48: A-CS | 0 | 0

80. Secondary Outcome: Treatment Phase 2 (Treatment Cycle 3)- Number of Participants With A-NCS and A-CS ECG Findings
Description: as for outcome 79
Time Frame: Week 12 and Week 48 (48 weeks after 1st treatment or withdrawal visit) in Treatment Cycle 3
Population: Safety Population 1. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
Number analyzed (Participants) | 5 | 3
Participants
  Week 12: A-NCS: number analyzed (Participants) | 4 | 2
  Week 12: A-NCS | 1 | 0
  Week 12: A-CS: number analyzed (Participants) | 4 | 2
  Week 12: A-CS | 0 | 0
  Week 48: A-NCS | 0 | 1
  Week 48: A-CS | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and Non-SAEs were collected up to 48 weeks in Treatment Cycle 1 and up to Week 48 (48 weeks after 1st treatment) in Treatment Cycles 2 and 3
Description: SAEs and non-SAEs were reported for SPDB Population (Treatment Cycle1:Placebo and GSK1358820 200 U) and Safety Population (SP) 1 (Treatment Cycle2:Placebo/GSK1358820 200 U), SP 2 (Treatment Cycle 2:GSK1358820 200 U/GSK1358820 200 U and Treatment Cycle 3: Placebo/GSK1358820 200 U) and SP 3 (Treatment Cycle3:GSK1358820 200 U/GSK1358820 200 U) .
Arm/Group | Treatment Cycle 1: Placebo | Treatment Cycle 1: GSK1358820 200U | Treatment Cycle 2: Placebo / GSK1358820 200 U | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U | Treatment Cycle 3: Placebo / GSK1358820 200 U | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11 | 0/10 | 0/6 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/11 | 1/10 | 0/6 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 5/10 | 8/11 | 5/10 | 5/6 | 4/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Cycle 1: Placebo (N=10) | Treatment Cycle 1: GSK1358820 200U (N=11) | Treatment Cycle 2: Placebo / GSK1358820 200 U (N=10) | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U (N=6) | Treatment Cycle 3: Placebo / GSK1358820 200 U (N=5) | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U (N=3)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Cycle 1: Placebo (N=10) | Treatment Cycle 1: GSK1358820 200U (N=11) | Treatment Cycle 2: Placebo / GSK1358820 200 U (N=10) | Treatment Cycle 2: GSK1358820 200 U / GSK1358820 200 U (N=6) | Treatment Cycle 3: Placebo / GSK1358820 200 U (N=5) | Treatment Cycle 3: GSK1358820 200 U / GSK1358820 200 U (N=3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3) | 3 (5) | 1 (1) | 2 (2) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasticity (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Occult blood (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/18/NCT02849418/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT02849418/SAP_001.pdf